CLINICAL TRIAL: NCT06343519
Title: Comparison of Echocardiographic and Laboratory Findings in Hemodynamic Monitoring of Shocked Patients
Brief Title: Echocardiographic and Laboratory Findings in Hemodynamic Monitoring of Shocked Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Atef Thabet Osman, Principal Investigator, Assiut University
Other Study IDs: Shocked Patients Monitoring
Record Dates: First submitted 2024-03-06; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Shock
MeSH Terms: conditions — Shock | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Echocardiography — Measuring echocardiographic parameters (cardiac index, speckle tracking, tissue Doppler indices)

SUMMARY:
Shocked patients require prompt and accurate assessment of their hemodynamic status to guide appropriate management. Echocardiography is a valuable tool for assessing cardiac function, while laboratory parameters such as mixed venous oxygen saturation and arterial blood lactate provide insights into tissue perfusion and oxygen metabolism. This study aims to compare echocardiographic findings, including cardiac index, speckle tracking parameters, and tissue Doppler indices, with laboratory findings in the evaluation of hemodynamic monitoring in shocked patients.

DETAILED DESCRIPTION:
Shocked individuals necessitate expeditious and precise evaluation of their hemodynamic condition to direct appropriate treatment. The utilization of echocardiography is an invaluable method for appraising cardiac function, while the inclusion of laboratory parameters such as mixed venous oxygen saturation and arterial blood lactate offers valuable insights into tissue perfusion and oxygen metabolism. The primary objective of this study is to compare the echocardiographic discoveries, which encompass the assessment of cardiac index, speckle tracking parameters, and tissue Doppler indices, with the laboratory findings in the comprehensive assessment of hemodynamic monitoring in individuals experiencing shock. The purpose of this investigation is to delineate the correlation between echocardiographic and laboratory assessments in order to enhance our understanding of hemodynamic status in patients who are in a state of shock.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with shock based on clinical criteria (e.g., hypotension, signs of tissue hypoperfusion) requiring hemodynamic monitoring.
* Patients age > 18 year old.

Exclusion Criteria:

* Patients with pre-existing cardiac conditions affecting echocardiographic parameters, those receiving mechanical circulatory support.
* Patients with contraindications to echocardiography or blood sampling.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients (age >18 years) presenting with shock admitted to the intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in Shock Status After Fluid Therapy Based on Echocardiographic Assessment of Fluid Responsiveness | 24 hours
  Change in shock status will be assessed 24 hours after initiation of fluid therapy by echocardiographic evaluation of cardiac index in liters per minute per square meter (L/min/m2).

CONTACTS AND LOCATIONS:
Overall Officials: Dina Ahmed, Study Director — Assiut University; Mohamed Maghraby, Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jardin F, Fourme T, Page B, Loubieres Y, Vieillard-Baron A, Beauchet A, Bourdarias JP. Persistent preload defect in severe sepsis despite fluid loading: A longitudinal echocardiographic study in patients with septic shock. Chest. 1999 Nov;116(5):1354-9. doi: 10.1378/chest.116.5.1354. PMID 10559099